CLINICAL TRIAL: NCT07261475
Title: Acute Effects of Water Extract of Crocus Sativus Tepals on Metabolic Health Parameters in Patients With Obesity and Prediabetes
Brief Title: Crocus Sativus Tepals Water Extract in Obesity and Prediabetes
Acronym: ZAFRAN
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Primorska (Other)
Collaborators: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Nina Mohorko, Associate professor, University of Primorska
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ZAFRAN-2025
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Prediabetes; Obesity & Overweight
Keywords: Crocus sativus tepals; Glycaemia; Oral glucose tolerance test; resting metabolism; blood pressure; insulin
MeSH Terms: conditions — Prediabetic State; Obesity; Overweight; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crocus sativus (Experimental): Crocus sativus tepals cold aqueous extract
  Interventions: Biological: Crocus sativus tepals cold aqueous extract
- water (Sham Comparator): cold water
  Interventions: Biological: cold water

INTERVENTIONS:
Biological: Crocus sativus tepals cold aqueous extract — 2 g of Crocus sativus tepals will be infused in 200 mL of water overnight at 4 °C, resulting cold aqueous extract corresponds to 40 mg GAE of polyphenols
  Arms: Crocus sativus
Biological: cold water — 200 mL of cold water, kept overnight at 4 °C
  Arms: water

SUMMARY:
The goal of this clinical trial is to determine the acute effects of ingestion of a cold aqueous extract of Crocus sativus tepals on postprandial glycemia and other indicators of metabolic health in patients with obesity and/or prediabetes. The main questions it aims to answer are:

* Does the ingestion of Crocus sativus tepals cold aqueous extract prior to a meal improve the glycemic response to a standard meal?
* How does the ingestion of Crocus sativus tepals aqueous extract prior to a meal impact insulin levels and other markers of metabolic health?
* Does the ingestion of Crocus sativus tepals cold aqueous extract prior to a meal increase the resting energy expanditure?

Researchers will compare Crocus sativus tepals cold aqueous extract to cold water.

The participants will visit the Faculty twice - on one visit they will ingest Crocus sativus tepals cold aqueous extract and on the other cold water (in random order) 5 minutes prior to a standard meal of 100 g of white bread.

On each visit, anthropometric measurements will be performed upon arrival. Blood samples will be collected 3 times, preceeded by resting metabolic rate and blood pressure measurements: at baseline in fasted conditions, and 60 minutes and 120 minutes after consuming the bread.

There will be an at least 7 days wash-out period between the two visits.

ELIGIBILITY:
Inclusion Criteria:

* Obesity type I (ITM > 30 kg/m2) and/or
* Prediabetes (fasting glucose levels 6,1 - 6,9 mmol/L)

Exclusion Criteria:

* Gastrointestinal diseases
* Diabetes mellitus of any type
* Pregnant or lactating, without contraception
* Serious clinical conditions such as cancer, severe infections, severe psychiatric disorders, autoimmune diseases, inflammatory diseases
* Participation in another clinical trial 3 months prior to the study
* ITM greater than 35 kg/m2
* Celiac disease of gluten intolerance
* electronic implant

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
glucose levels | From enrollment to the end of second measurement at 2 weeks
  Serum glucose levels will be measured from venous blood at baseline and 60 and 120 minutes after bread ingestion.

SECONDARY OUTCOMES:
insulin level | From enrollment to the end of second measurement at 2 weeks.
  Serum insulin levels will be measured from venous blood at baseline and 60 and 120 minutes after bread ingestion.
Resting metabolism | From enrollment to the end of the second measurement, at 2 weeks
  Resting metabolism will be measured with indirect calorimetry at baseline in fasted state and at 40 and 100 minutes after bread ingestion.
  To determine RMR, subjects will lie relaxed on a bed in a thermoneutral room for 10 minutes to calm down, followed by a 20-minute measurement of oxygen consumption (VO2) and carbon dioxide production (VCO2). RMR and RQ will be calculated from stable values over a 15-minute period (the first 5 minutes of measurement until stabilization will not be taken into account).
Blood pressure | baseline, 60 minutes after bread ingestion, 120 minutes after bread ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Nina Mohorko, PhD, Principal Investigator — University pf Primorska, Faculty of Health Sciences
Locations (1):
- University pf Primorska, Faculty of Health Sciences, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barik SK, Sengupta S, Arya R, Kumar S, Kim JJ, Chaurasia R. Dietary Polyphenols as Potential Therapeutic Agents in Type 2 Diabetes Management: Advances and Opportunities. Adv Nutr. 2025 Jan;16(1):100346. doi: 10.1016/j.advnut.2024.100346. Epub 2024 Nov 19. PMID 39566886
- [Background] Omidi A, Riahinia N, Montazer Torbati MB, Behdani MA. Hepatoprotective effect of Crocus sativus (saffron) petals extract against acetaminophen toxicity in male Wistar rats. Avicenna J Phytomed. 2014 Sep;4(5):330-6. PMID 25386395
- [Background] Moratalla-Lopez N, Bagur MJ, Lorenzo C, Salinas MEMR, Alonso GL. Bioactivity and Bioavailability of the Major Metabolites of Crocus sativus L. Flower. Molecules. 2019 Aug 2;24(15):2827. doi: 10.3390/molecules24152827. PMID 31382514
- [Background] Montoro P, Maldini M, Luciani L, Tuberoso CI, Congiu F, Pizza C. Radical scavenging activity and LC-MS metabolic profiling of petals, stamens, and flowers of Crocus sativus L. J Food Sci. 2012 Aug;77(8):C893-900. doi: 10.1111/j.1750-3841.2012.02803.x. Epub 2012 Jul 18. PMID 22809329
- [Background] Menghini L, Leporini L, Vecchiotti G, Locatelli M, Carradori S, Ferrante C, Zengin G, Recinella L, Chiavaroli A, Leone S, Brunetti L, Orlando G. Crocus sativus L. stigmas and byproducts: Qualitative fingerprint, antioxidant potentials and enzyme inhibitory activities. Food Res Int. 2018 Jul;109:91-98. doi: 10.1016/j.foodres.2018.04.028. Epub 2018 Apr 16. PMID 29803496
- [Background] Bursac B, Bellachioma L, Gligorovska L, Jovanovic M, Teofilovic A, Vrataric M, Vojnovic Milutinovic D, Albacete A, Martinez-Melgarejo PA, Morresi C, Damiani E, Bacchetti T, Djordjevic A. Crocus sativus tepals extract suppresses subcutaneous adipose tissue hypertrophy and improves systemic insulin sensitivity in mice on high-fat diet. Biofactors. 2024 Jul-Aug;50(4):828-844. doi: 10.1002/biof.2043. Epub 2024 Feb 6. PMID 38318672
- [Background] Bellachioma L, Morresi C, Albacete A, Martinez-Melgarejo PA, Ferretti G, Giorgini G, Galeazzi R, Damiani E, Bacchetti T. Insights on the Hypoglycemic Potential of Crocus sativus Tepal Polyphenols: An In Vitro and In Silico Study. Int J Mol Sci. 2023 May 24;24(11):9213. doi: 10.3390/ijms24119213. PMID 37298165